CLINICAL TRIAL: NCT01586546
Title: Quality of Life Outcomes Following Mind-body Skills Training for Cancer Patients That Are Facilitated Either Face-to-face or Online: A Pilot Study
Brief Title: A Pilot Study To Assess Guidance in and Subsequent Use of Mind-Body Techniques on the Quality of Life of Cancer Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Encountered significant recruitment challenges, and it was decided to terminate the study without recruiting participants.
Sponsor: Absenger Cancer Education Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MBM 5538
Record Dates: First submitted 2012-04-23; First posted 2012-04-27 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Quality of Life; Life Change Events; Neoplasms
Keywords: Mind-body; Psychosocial; Meditation; Breathing Exercises; Guided Imagery; Visualization
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Face-to-Face MBM Skills Group (Experimental)
  Interventions: Behavioral: Face-to-Face MBM Skills Group
- Online MBM Skills Group (Experimental)
  Interventions: Behavioral: Online MBM Skills Group
- Waitlist Control I (Other): This group will be given the option to participate in a face-to-face MBM skills group intervention after conclusion of study.
  Interventions: Other: Waitlist Control I
- Waitlisted Control II (Other): This group will be given the option to participate in an Online MBM skills group intervention after conclusion of study.
  Interventions: Other: Waitlist Control II

INTERVENTIONS:
Behavioral: Face-to-Face MBM Skills Group — Mind Body Medicine (MBM) Skills Groups provide a means for study participants to learn skills for taking care of themselves in a supportive small group setting. Participants will learn and practice a variety of specific MBM skills. These MBM skills will enable a participant to change the way she/he deals with the wide range of stressors at different stages of her/his cancer journey. Some of these MBM skills are meditation, guided imagery, biofeedback, writing, and drawing. These groups are designed to assist a participant in coming to know themselves better and in learning and using these tools that will help the participant to deal with the distress as only a small percentage of cancer patients in distress receive appropriate support.
  Arms: Face-to-Face MBM Skills Group
Other: Waitlist Control I — No intervention offered during study period. Intervention is offered after completion of study.
  Arms: Waitlist Control I
Other: Waitlist Control II — No intervention offered during study period. Intervention is offered after completion of study.
  Arms: Waitlisted Control II
Behavioral: Online MBM Skills Group — Mind Body Medicine (MBM) Skills Groups provide a means for study participants to learn skills for taking care of themselves in a supportive small group setting. Participants will learn and practice a variety of specific MBM skills. These MBM skills will enable a participant to change the way she/he deals with the wide range of stressors at different stages of her/his cancer journey. Some of these MBM skills are meditation, guided imagery, biofeedback, writing, and drawing. These groups are designed to assist a participant in coming to know themselves better and in learning and using these tools that will help the participant to deal with the distress as only a small percentage of cancer patients in distress receive appropriate support.
  Arms: Online MBM Skills Group

SUMMARY:
Aim: To answer the questions of whether a Mind-Body Medicine (MBM) skills group facilitated face-to-face and online can improve measures of Quality of Life (QOL) in a population of cancer patients.

Value of Study: Technological advances have contributed to new venues for healthcare delivery. It is imperative that these new delivery methods, for individual and/or group psychosocial services are sufficiently tested and validated. Research shows that there is very little knowledge about differences in communication styles between online and face-to-face groups, nor is there much knowledge on the overall efficacy of online groups.

Phenomenon Studied: Can MBM skills groups improve the quality of life of cancer patients? Is there a difference in outcome between a MBM skills group delivered face-to-face and a MBM skills group delivered online.

Reasons Leading to Proposing the Project: Despite encouraging research showing that psychosocial interventions have positive effects in the lives of cancer patients, more research is needed due to several problems of current research, such as poor study design, lack of use of technological advances and relatively few existing studies on the effectiveness of MBM therapies in the oncological setting.

Stated Hypothesis:

Hypothesis 1:

There is no difference between baseline QOL measures and QOL measures at the end of face-to-face facilitated MBM skills groups.

Hypothesis 2:

There is no difference between baseline QOL measures and QOL measures at the end of Online facilitated MBM skills groups.

Hypothesis 3:

Participation in either, online facilitated MBM skills groups or face-to-face facilitated MBM skills groups will improve QOL measures when compared to control group.

Hypothesis 4:

Patients in the control group (waitlist control, care as usual group) will have no improvement on QOL measures.

Anticipated Value to the Larger Community: According to the National Center for Complementary and Alternative Medicine (NCCAM) "…there is a need for reliable, objective, evidence-based information regarding the usefulness and safety-or lack thereof-of CAM" (National Center for Complementary and Alternative Medicine, 2011, p.3). This study will add to general scientific knowledge of CAM and MBM.

ELIGIBILITY:
Inclusion Criteria:

* TNM staged tumors Stage I to Stage IV,
* Tumors staged according to the Ann Arbor staging classification system (commonly lymphomas)
* Tumors which don't have a clear-cut staging system such as most types of leukemia and blood or bone marrow cancers
* Tumors staged by the International Federation of Gynecology and Obstetrics (cervix, uterus, ovary, vagina, and vulva).
* No neurological illness

Exclusion Criteria:

* Mental functioning clinically estimated to be below the low average range (IQ< 80). (Impaired cognitive level might impede verbal comprehension).
* Not being able to speak or understand English;
* No access to reliable computer with operational software to participate in online video conferences
* Unavailability of built-in or external web-cam
* Unavailability of reliable high-speed Internet connection
* Unavailability of reliable transportation to and from face-to-face MBM skills group meetings
* Barring unforeseen circumstances, intent to participate in each and every one of the eight MBM Skills Groups session

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Quality Of Life, as assessed by the World Health Organization Quality of Life (WHOQOL-BREF) instrument | Baseline, week 4
  The WHOQOL-BREF is a 26-item version of the WHOQOL-100 assessment. The instrument has been tested and developed for almost 20 years and "…results indicate that overall, the WHOQOL-BREF is a sound, cross-culturally valid assessment of QOL, as reflected by its four domains: physical, psychological, social and environment" (Skevington, Lofty, & O'Connell, 2004).

SECONDARY OUTCOMES:
Change in distress, anxiety, depression and need for help as assessed by the Emotion Thermometers Tool© (ET5) | Baseline, Week 4
  The ET5 is a five dimensional tool comprised of five visual-analogue scales in the form of four predictor domains (distress, anxiety, depression, anger) and one outcome domain (need for help). It is modeled after the original Distress Thermometer (DT) recommended by the US National Comprehensive Cancer Network. In order to detect broadly defined distress or anxiety, a combination of thermometers was most accurate (Mitchell, Baker-Glenn, Park, Granger, & Symonds, 2010). The ET5 tool expands on the DT by combining domains in order to detect emotional complications after a diagnosis with cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Werner Absenger, M.Sc., Principal Investigator — Absenger Cancer Education Foundation, Spring Lake, Michigan & Saybrook University's College of Mind-Body Medicine, San Francisco, California
Locations (1):
- Absenger Cancer Education Foundation, Spring Lake, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Absenger Cancer Education Foundation Homepage — http://amacf.org